CLINICAL TRIAL: NCT06730594
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Design Clinical Study to Assess the Effect of the Bio-K+ Probiotic Capsules (VL-BK-02) in Adults With Functional Constipation
Brief Title: A Study to Assess the Effect of the Bio-K+ Probiotic Capsules (VL-BK-02) in Adults With Functional Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KE/240401/BK+/FC
Record Dates: First submitted 2024-11-13; First posted 2024-12-12 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-01

CONDITIONS: Functional Constipation
MeSH Terms: interventions — microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Parallel Assignment A randomized, double-blind, two-arm, placebo-controlled clinical study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VL-BK-02 (25 billion CFU/Capsule) (Experimental): One capsule per day to be consumed orally before breakfast Duration: 84 days (12 weeks)
  Interventions: Dietary Supplement: VL-BK-02 (25 billion CFU/Capsule)
- Placebo (Microcrystalline Cellulose - 375 mg/capsule) (Placebo Comparator): One capsule per day to be consumed orally before breakfast Duration: 84 days (12 weeks)
  Interventions: Dietary Supplement: Placebo (Microcrystalline Cellulose - 375 mg/capsule)

INTERVENTIONS:
Dietary Supplement: VL-BK-02 (25 billion CFU/Capsule) — One capsule per day consumed orally before breakfast Duration: 84 days (12 weeks)
  Arms: VL-BK-02 (25 billion CFU/Capsule)
Dietary Supplement: Placebo (Microcrystalline Cellulose - 375 mg/capsule) — One capsule per day consumed orally before breakfast Duration: 84 days (12 weeks)
  Arms: Placebo (Microcrystalline Cellulose - 375 mg/capsule)

SUMMARY:
The present study is a randomized, placebo-controlled, double-blind, parallel-group clinical study designed to assess the effects of IP in individuals with Functional constipation as compared to a placebo. Approximately 205 individuals aged between 18 and 60 years will be screened.

Considering a screen failure of 20%, approximately 164 individuals will be randomized in a ratio of 1:1 to receive either the active or placebo. The study will have at least 126 completed participants i.e. 63 partcipants in each study arm after accounting for a dropout/withdrawal rate of 23% at the end of the study. The intervention duration for all the study participants will be 56 days with follow up of upto 84 days. The study flow chart given below indicates the time points at which safety and efficacy assessments will be conducted

ELIGIBILITY:
Inclusion Criteria:

1. Individuals agreed to the signed and dated informed consent form.
2. Male and female individuals of age between 18 to 60 years (both values included)
3. Individuals who meet Rome IV diagnostic criteria for functional constipation is indicated by the following criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis:

   i. Fewer than three SBM per week ii. Any one or more of the below criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis:
   1. Straining during more than ¼ (25%) of defecations
   2. Lumpy or hard stools (Bristol Stool Form Scale 1-2) more than ¼ (25%) of defecations
   3. Sensation of incomplete evacuation more than ¼ (25%) of defecations
   4. Sensation of anorectal obstruction/ blockage more than ¼ (25%) of defecations
   5. Manual maneuvers to facilitate more than ¼ (25%) of defecations (e.g., digital evacuation, support of the pelvic floor) iii. Loose stools are rarely present without the use of laxatives iv. Insufficient criteria for irritable bowel syndrome
4. Individuals willing to comply with all study procedures and availability for the duration of the study as per the protocol.
5. Individuals willing to maintain the same dietary and physical activity practices throughout the study period.

Exclusion Criteria:

1. Individuals with well-known, organic causes of constipation (Polyps, hemorrhoids, etc.)
2. Individuals with anorectal pathology
3. Individuals with a history of previous gastrointestinal surgery.
4. Individuals with any alarming symptoms (i.e. rectal bleeding, weight loss, jaundice) as judged by the Investigator.
5. Individuals with concurrent chronic GI pathology (e.g. IBD, cystic fibrosis, short gut, celiac disease, food allergy, Frequent diarrhea without laxatives).
6. Current pharmacological treatment related to constipation (e.g. prosecretory agents, antibiotics, antidepressants, antispasmodics, enterokinetic)
7. Individuals consuming dietary treatment (e.g. synbiotics, herbal extracts, fibers) or taking other therapies for treating constipation (e.g. cognitive behavior therapy, acupuncture, biofeedback, complementary and alternative Medicine) within 1 month prior to screening.
8. Use of antibiotics within 1 month prior to screening
9. Use of products containing probiotics within 1 month prior to screening
10. Opioids-induced constipation
11. Regular use of any drug or dietary supplement known to cause constipation (e.g. iron, opioids, sucralfate, misoprostol, 5-HT- antagonists, antacids with magnesium, calcium or aluminum, antidiarrheal medication, anticholinergic agents, calcium supplements, calcium channel blockers, tricyclic antidepressants or NSAIDs) within 1 month before the screening.
12. Immuno-compromised participants or those on immunosuppressive agents (e.g. heart or kidney transplant, chemotherapy agents, oral prednisolone)
13. History of cancer.
14. Individuals with known history of diabetes mellitus and are on medication for the same.
15. History of uncontrolled hypertension and/or systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg.
16. Individuals with impaired thyroid function reported by TSH less than 0.4 mIU/L and more than 5 mIU/L will be excluded. However, individuals on a stable dose of medication for past 6 months and within the aforementioned range, can be considered.
17. Mental or behavioral disorders as judged by the Investigator.
18. Individuals with known food allergy.
19. Individuals with eating disorders (e.g., anorexia, bulimia).
20. Pregnancy or lactation.
21. Known allergic reactions to any components of the probiotics or placebo.
22. Individuals participating in other interventional study within 90 Days prior to screening.
23. Individuals with a history of alcohol or drug abuse based on medical history, physical examination, or the Investigators clinical judgment.
24. Current Smokers will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of VL-BK-02 on changes in the frequency of Complete Spontaneous Bowel Movements (CSBMs) | per week from baseline to the end of study visit.
  Severe constipation is defined as no complete spontaneous bowel movements (CSBMs) and an average straining score ≥ 3.0 (CIC; 5-point scale) CSBM has emerged as an attractive symptom-specific primary endpoint for constipation trials, as it integrates the objective, quantitative sign of stool frequency and the subjective, qualitative symptom of sensation of complete defecation

SECONDARY OUTCOMES:
To assess the effect of Investigational product (IP) in comparison to baseline and placebo on Stool consistency as assessed by Bristol Stool Form Scale (BSFS) | Baseline to Day 84
  The BSFS is a commonly used ordinal stool-type scale in clinical research and practice that goes from the hardest (type 1) to the softest (type 7). Abnormally hard stools (and in conjunction with other symptoms indicative of constipation) are referred to as types 1 and 2. On the other hand, types 6 and 7 are characterized by unusually loose or watery stools together with other symptoms that point to diarrhea. Stool forms 3-5 are regarded as the most "normal.
To assess the effect of Investigational product (IP) in comparison to baseline and placebo on Constipation symptoms by using Participant Assessment of Constipation Symptoms (PAC-SYM) | Baseline to day 14, day 28, day 42, day 56, day 70 and day 84.
  Chronic constipation is a common, self-reported, symptom-based disorder, which can significantly impact an individual's health-related quality of life The 12-item questionnaire is divided into three symptom subscales: abdominal (four items); rectal (three items); and stool (five items). Items are scored on 5-point Likert scales, with scores ranging from 0 to 4 (0 = 'symptom absent', 1 = 'mild', 2 = 'moderate', 3 = 'severe', and 4 = 'very severe'). A mean total score in the range of 0-4 is generated by dividing the total score by the number of questions completed; the lower the total score, the lower the symptom burden.
To assess the effect of Investigational product (IP) in comparison to baseline and placebo on Quality of life by using Participant Assessment of Constipation QoL (PAC-QoL) | Baseline to day 14, day 28, day 42, day 56, day 70 and day 84.
  The PAC-QOL questionnaire is subcategorized into 4 items on physical discomfort, 8 items on psychosocial discomfort, 5 items on treatment satisfaction, and finally 11 items on worries and discomfort. Response choice is a Likert scale from 0 to 4.Higher scores mean higher negative effects on quality of life. Items
To assess the effect of Investigational product (IP) in comparison to baseline and placebo Percentage responders are defined as the number of participants with an increase by 1 or more frequencies of SBM with no sensation of incomplete evacuation | Baseline to Day 84
  A spontaneous bowel movement (SBM) is defined as a stool passed spontaneously without induction by any medication and a CSBM is defined as an SBM with a sensation of complete evacuation
To assess the effect of Investigational product (IP) in comparison to baseline and placebo Gut microbiome (alpha and beta diversity) | Baseline to Day 84
  Stool samples will be collected from the participants on Day 0 and Day 56. A window period of ± 3 days will be provided for stool sample collection. Participants will be provided with a stool sample collection kit with sample collection instructions on screening day and day 28. Stool samples will be collected from participants's homes or on site at Day 0 and Day 56. The samples will be further stored for future analysis of metagenome NGS sequencing. Stool samples will be collected from the participants and shipped to the central lab in gel ice pack. Stool samples for NGS will be stored at -80 degrees until shipped to the central lab
To assess the effect of Investigational product (IP) in comparison to baseline and placebo Difference in the usage of rescue medication throughout the study duration as compared to placebo. | through study completion, an average of Day 84
  Bowel movement within 24 hours of consuming the rescue medication will not be considered as an SBM or a CSBM

CONTACTS AND LOCATIONS:
Locations (8):
- India (8):
  - Anand Multispeciality Hospital, Vadodara, Gujarat
  - HCG Hospitals, Ahmedabad, Gujrata
  - Jan Kalyan Multispeciality Hospital, Kalyān, Maharashtra
  - Signus Hospital, Nashik, Maharashtra
  - AK Superspeciality Clinic, Pune, Maharashtra
  - Lifeline multispecialty Hospital, Pune, Maharashtra
  - Care Multispecialty Hospital, Pune, Maharashtra
  - Krishna Hospital, Varanasi, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No